CLINICAL TRIAL: NCT06344520
Title: The Effect of Minor Muscle Stretching Exercises on the Motor Control and Swimming Speed of Young Swimmers
Brief Title: Pectoralis Minor Shorthening and Swimming Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Dilan Siriş, physiotheraepist, Istinye University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IsiU
Record Dates: First submitted 2024-03-20; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: The Study Will Not be Based on Any Disease; Ability to Swim 100m Independent Freestyle; Be Between the Ages of 9-16; Continuing Running as Part of a Sports Club
Keywords: Swimmers; pectoralis minör
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: three groups as intervention, exercises group non- exercises group and scham
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pectoralis minor stretching exercise group (Experimental): They observed the effects of shoulder stabilization exercises and pectoralis minor stretching exercises on balance and maximal shoulder strength in their study on healthy young people with rounded shoulder posture. Based on this, the pectoralis minor stretching exercise to be performed in swimmers not only corrects the maldeveloped posture in children, but also increases maximal shoulder muscle strength. It is aimed to increase swimming performance by contributing to the increase in swimming performance.Volunteer athletes who agreed to participate in the thesis were initially administered tests measuring balance, posture, motor control and swimming speed. After the tests, in addition to their own training, 3 pectoralis minor stretching exercises with a total duration of 15 minutes, as specified by Mi-Kyoung et al. (2018), were applied for 8 weeks, at least 2 times a week.
  Interventions: Behavioral: pektoralis minor shortnes
- Group in which the sham Pectoralis Minor stretching exercise (Sham Comparator): Volunteer athletes who agreed to participate in the thesis were initially administered tests measuring balance, posture, motor control and swimming speed. After the tests, in addition to their own training, 3 sham pectoralis minor stretching exercises with a total duration of 15 minutes, were applied for 8 weeks, at least 2 times a week.
  Interventions: Behavioral: Group in which the Pectoralis Minor stretching exercise was performed in a sham manner
- The group in which Pectoralis Minor stretching exercise was not applied (Active Comparator): Volunteer athletes who agreed to participate in the thesis were initially administered tests measuring balance, posture, motor control and swimming speed. After the tests,They continued to do their own training
  Interventions: Behavioral: The group in which Pectoralis Minor stretching exercise was not applied

INTERVENTIONS:
Behavioral: pektoralis minor shortnes — One factor that is effective in acceleration during swimming is the force of the arm pulling the water. While the pectoralis minor muscle pulls the crocoid process forward, it pulls its posterolateral corner down, which helps the latismus dorsi to make an extension movement and the lower trapezius to depress the scapula. When the pectoralis minor muscle is short, it prevents maximum reach in the arm because its full function cannot be revealed. It is thought that depression of the scapula will directly affect acceleration in swimming, as it increases the backward thrust of the arm.
  Arms: Pectoralis minor stretching exercise group
Behavioral: Group in which the Pectoralis Minor stretching exercise was performed in a sham manner — In most cases, exercise practices also affect the person psychologically. In order to ignore the psychological effects of the exercises, they were made to perform exercises that were similar to pectoralis minor stretching exercises but did not activate the muscle
  Arms: Group in which the sham Pectoralis Minor stretching exercise
Behavioral: The group in which Pectoralis Minor stretching exercise was not applied — The Control Group was not given any exercise and they continued to do their own training.
  Arms: The group in which Pectoralis Minor stretching exercise was not applied

SUMMARY:
Swimming is one of the sports branches that includes many factors such as aerobic and anaerobic endurance, strength, flexibility, speed, quickness, rhythm, coordination as well as sportive performance and technical skills.

Athletes must have a high level of fitness, strength, coordination, agility, speed and motor control to perform at an elite level with minimal injury risk.

Repetitive upper extremity movements imposed by freestyle swimming may lead to changes in muscle length and tension by paving the way for postural misalignment in adolescent swimmers.

As can be seen in the studies, young swimmers who are preparing for the competition have postural disorders and injuries related to use, such as decreased posture, shoulder joint range of motion and subacromial distance.

Pectoralis minor stretching exercise to be performed in swimmers is aimed to improve swimming performance and prevent possible postural disorders by contributing to the increase of maximal shoulder muscle strength as well as correcting the incorrectly developed posture in children.

DETAILED DESCRIPTION:
Sport has become a necessity for a healthy and balanced life today. Children who play sports regularly at a young age become adults who do sports later in their lives. Swimming is one of the sports branches that includes many factors such as aerobic and anaerobic endurance, strength, flexibility, speed, quickness, rhythm, coordination as well as sportive performance and technical skills. Swimming is not only a sport, but also provides a symmetrical and balanced development of some muscles as well as making use of free time, gaining strength and rehabilitation.

The primary function of the nervous system in all living things is movement. Parallel to the phylogenetic development, there is also an improvement in the movement function. The realization of a movement is not possible only with the operation of the pyramidal system, which is the primary movement system. In addition, the extrapyramidal system that will provide the most appropriate postural tone for the organ that will perform the voluntary movement towards the goal, the cerebellar system that will provide the coordination of the agonist antagonist muscles, and the awake state must be normal and the level of consciousness must be open for this movement. The sum of the systems that provide all this movement is called the motor system. The factor that ensures the harmonious operation of the movement emerging from this system is motor control.

Athletes must have a high level of fitness, strength, coordination, agility, speed and motor control to perform at an elite level with minimal injury risk. Dysfunctional movement patterns are directly related to the mechanism of injury. In addition, the improvement of motor control is directly related to the prevention of injury. It is very important to prevent injury in order to ensure continuity in sports in athletes.

Repetitive upper extremity movements imposed by freestyle swimming may lead to changes in muscle length and tension by paving the way for postural misalignment in adolescent swimmers . Study, revealed that there were great differences in sagittal stance angles of freestyle swimming female adolescent athletes compared to their non-swimming peers, and adolescent athletes engaged in swimming sports had far from the desired angles in sagial stance.

One of the parameters affecting swimming sport is muscle strength. While four techniques are used as freestyle, backstroke, breaststroke and butterfly, swimming speed is considered to be the most important performance indicator in all. Swimming speed is defined as completing the 25m or 50m swimming distance in the pool in the shortest time and is considered the most important feature of the swimmer that needs to be developed in terms of trainers. Lower extremity strength is also accepted as an important criterion in terms of starting swimming and especially completing the first 15 meters .

Intrinsic and extrinsic factors are effective in the prevention of acute, subacute and chronic injuries in sports . The most important system affecting these intrinsic and extrinsic factors is the Sensorymotor system. The sensorymotor system, on the other hand, is defined as the system that provides sensory, motor and central integration to ensure functional joint stability. Swimming; It is a sport branch that includes many factors such as high level aerobic and anaerobic endurance, strength, flexibility, speed, quickness, rhythm, coordination, sportive performance and technical skills .

As can be seen in the studies, young swimmers who are preparing for the competition have postural disorders and injuries related to use, such as decreased posture, shoulder joint range of motion and subracromial distance. In this context, it is important to see the effects of the studies applied on land and motor control on the performance in water and to ensure that the deficiencies are eliminated. As with any sport, swimming is a sport with a risk of injury. The presence of asymmetry between general leg strength, which is also observed among elite athletes, will negatively affect performance. An effective factor in acceleration during swimming is the force of the arm while pulling the water. The lower trapezius, latismus dorsi, pectoralis minor, and the supclavius muscle work as the scapula-thoracic depressor. The lower trapezius and pectoralis minor muscles directly affect the scapula, while the latismus dorsi muscle helps by pushing the humerus inferiorly. While the pectoralis minor muscle pulls the crocoid process forward, it lowers its posterolateral corner, which helps the latismus dorsi to extend and the lower trapezius to depress the scapula. In the shortness of the pectoralis minor muscle, the full function cannot be revealed, thus preventing the maximum extension of the arm. The shortness of the pectoralis minor muscle causes a postural disorder called the round shoulder. It is important to increase the mobility of the shoulder by stretching this muscle in terms of the smoothness of the posture. Since the depressed scapula increases the backward thrust of the arm, it is thought that it will directly affect the acceleration in swimming sports. They observed the effects of shoulder stabilization exercises and pectoralis minor stretching exercises on balance and maximal shoulder strength in a study conducted on healthy young people with a rounded shoulder posture. Based on these, pectoralis minor stretching exercise to be performed in swimmers is aimed to improve swimming performance and prevent possible postural disorders by contributing to the increase of maximal shoulder muscle strength as well as correcting the incorrectly developed posture in children.

ELIGIBILITY:
Inclusion Criteria:

* Ability to swim 100m independent freestyle
* Be between the ages of 9-16
* Continuing running as part of a sports club

Exclusion Criteria:

* Not accepting to work
* Injury history in the last 3 months
* Having received physiotherapy in the last 6 months
* Having a systemic disorder

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Speed Tests | 2 Mounths
  Swimming Speed: The Swimming Speed Of Children And Young People Preparing For The Competition Will Be Measured With A Stopwatch By An Experienced Coach.
Apley test | 2 Mounths
  The test is performed by looking at the distance of the arm to be tested from the crossed scapula. External rotation and abduction of the arm are checked.
  Shoulder protraction measurement: While the participants are in a comfortable position with their backs against the wall, the position of the shoulder is measured by measuring the distance from the front end of the acromion to the wall.
Round Shoulder | 2 Mounth
  For shoulder protraction (round shoulder) measurement, the position of the shoulder is measured by measuring the distance from the front end of the acromion to the wall while the participants are in a comfortable position with their backs against the wall. The protraction of the shoulder is determined by determining the distance from the anterior end of the acromion, which should normally be in contact with the wall, to the wall.
Anthropometric Measurement: | 2 Mounth
  Body Mass Index : The mesurment is in kg/m^2
Posture analysis: (ANNEX2) | 2 Mounth
  Posture analysis: (ANNEX2) It will be measured with the New York Posture analysis test. NYP.The highest score is 65 and the lowest score is 0. It is a scale that shows that the higher the score, the better the person's posture.
Anthropometric Measurement 2 | 2 Mounth
  Fathom Measurement: The Participant Leans On The Scale With His Arms : the measurment is in meters
Y Balance Test | 2 Mounth
  Y Balance Test is a test that is suitable for use in many different sports branches and evaluates lower extremity functional movement capacity, balance and motor control
Eurofit Test Battery | 2 Mounth
  Strength Tests : Hand strength will be measured in kilograms with a hand dynameter.
Eurofit Test Battery 2 | 2 Mounth
  Flexibility Tests:In the flexibility test, the distance the person can reach forward while sitting on the floor with his legs straight will be measured in centimeters.
Eurofit Test Battery 3 | 2 Mounth
  Sit-Up Test : The person lies on the ground on his back with his knees bent and puts his arms behind his head. The stopwatch is kept for 30 seconds while the number of times the person lifts his back from the ground, approaches his feet and lies down again is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Habibe Serap İnal, PhD, Study Director — İstinye Univercity
Locations (1):
- Galatasaray Ergün Gürsoy Olympic Swimming Pool, Üsküdar, Nuhkuyusu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The effects of shoulder stabilization exercises and pectoralis minor stretching on balance and maximal shoulder muscle strength of healthy young adults with round shoulder posture — https://pubmed.ncbi.nlm.nih.gov/29581654/
- Available data/document: Clinical Study Report — https://pubmed.ncbi.nlm.nih.gov/33842036/ — Athletes must have a high level of fitness, strength, coordination, agility, speed and motor control to perform at an elite level with minimal injury risk
- Available data/document: Clinical Study Report — https://pubmed.ncbi.nlm.nih.gov/22607780/ — Dysfunctional movement patterns are directly related to the mechanism of injury
- Available data/document: Clinical Study Report — https://pubmed.ncbi.nlm.nih.gov/27215935/ — In addition, the improvement of motor control is directly related to the prevention of injury
- Available data/document: Clinical Study Report — https://acikerisim.gelisim.edu.tr/xmlui/handle/11363/323 — Sport has become a necessity for a healthy and balanced life today. Children who play sports regularly at a young age become adults who do sports later in their lives. Swimming is one of the sports branches that includes many factors such as aerobic and anaerobic endurance, strength, flexibility, speed, quickness, rhythm, coordination as well as sportive performance and technical skills. Swimming is not only a sport, but also provides a symmetrical and balanced development of some muscles as well as making use of free time, gaining strength and rehabilitation.
- Available data/document: Clinical Study Report — https://www.researchgate.net/publication/356845509_Comparative_upper-quarter_posture_analysis_of_female_adolescent_freestyle_swimmers_and_non-swimmers — Repetitive upper extremity movements imposed by freestyle swimming may lead to changes in muscle length and tension by paving the way for postural misalignment in adolescent swimmers . Botha et al. (2022), in their study, revealed that there were great differences in sagittal stance angles of freestyle swimming female adolescent athletes compared to their non-swimming peers, and adolescent athletes engaged in swimming sports had far from the desired angles in sagial stance
- Available data/document: Clinical Study Report — https://research.usc.edu.au/esploro/outputs/99449442202621 — One of the parameters affecting swimming sport is muscle strength. While four techniques are used as freestyle, backstroke, breaststroke and butterfly, swimming speed is considered to be the most important performance indicator in all
- Available data/document: Clinical Study Report — https://pubmed.ncbi.nlm.nih.gov/20664366/ — Lower extremity strength is also accepted as an important criterion in terms of starting swimming and especially completing the first 15 meters
- Available data/document: Clinical Study Report — https://pubmed.ncbi.nlm.nih.gov/20699426/ — Intrinsic and extrinsic factors are effective in the prevention of acute, subacute and chronic injuries in sports
- Available data/document: Clinical Study Report — https://pubmed.ncbi.nlm.nih.gov/19442581/ — The sensorymotor system, on the other hand, is defined as the system that provides sensory, motor and central integration to ensure functional joint stability
- Available data/document: Clinical Study Report — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC164311/ — Swimming; It is a sport branch that includes many factors such as high level aerobic and anaerobic endurance, strength, flexibility, speed, quickness, rhythm, coordination, sportive performance and technical skills
- Available data/document: Clinical Study Report — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4851131/ — As can be seen in the studies, young swimmers who are preparing for the competition have postural disorders and injuries related to use, such as decreased posture, shoulder joint range of motion and subacromial distance
- Available data/document: Clinical Study Report — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5857441/ — Mi-Kyoung et al. (2018) observed the effects of shoulder stabilization exercises and pectoralis minor stretching exercises on balance and maximal shoulder strength in a study conducted on healthy young people with a rounded shoulder posture.
- Available data/document: Book: D.A. Neumann, — https://shop.elsevier.com/books/kinesiology-of-the-musculoskeletal-system/neumann/978-0-323-28753-1 — An effective factor in acceleration during swimming is the force of the arm while pulling the water. The lower trapezius, latismus dorsi pectoralis minor, and the supclavius muscle work as the scapula-thoracic depressor. The lower trapezius and pectoralis minor muscles directly affect the scapula, while the latismus dorsi muscle helps by pushing the humerus inferiorly. While the pectoralis minor muscle pulls the crocoid process forward, it lowers its posterolateral corner, which helps the latismus dorsi to extend and the lower trapezius to depress the scapula
- Available data/document: Clinical Study Report — https://pubmed.ncbi.nlm.nih.gov/14573714/ — In the shortness of the pectoralis minor muscle, the full function cannot be revealed, thus preventing the maximum extension of the arm. The shortness of the pectoralis minor muscle causes a postural disorder called the round shoulder. It is important to increase the mobility of the shoulder by stretching this muscle in terms of the smoothness of the posture. Since the depressed scapula increases the backward thrust of the arm, it is thought that it will directly affect the acceleration in swimming sports